CLINICAL TRIAL: NCT03514914
Title: Enhancing Male Participation in Interventions to Prevent Unintended Pregnancy
Acronym: CHARM2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Population Council (Other)
Responsible Party: Principal Investigator, Anita Raj, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1R01HD084453-01A1 (NIH)
Record Dates: First submitted 2018-04-10; First posted 2018-05-03 (Actual); Results first posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: Contraception
Keywords: LARC, contraception, family planning, India, male engagement

STUDY DESIGN:
Intervention Model Description: To evaluate the impact of CHARM2 on reversible contraceptive use (including LARC), unintended pregnancy, and MSV via a two armed cluster RCT with N=1000-1200 married couples from 20 geographic clusters (n=50-60 couples per cluster) in rural India. The control arm will receive standard of care in the form of community health workers offering pills/condoms and linking women to public health clinics.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHARM2 Intervention (Experimental): CHARM2 intervention will involve gender, culture & contextually-tailored family planning and gender equity counseling for married couples. Two sessions for men delivered by male health providers and two sessions for women delivered by female providers.
  Interventions: Behavioral: The CHARM2 Intervention
- Control (No Intervention): Control clusters will receive standard of care.

INTERVENTIONS:
Behavioral: The CHARM2 Intervention — CHARM2 intervention will involve gender, culture & contextually-tailored family planning and gender equity counseling.
  Arms: CHARM2 Intervention

SUMMARY:
Globally, 41% of all pregnancies are unintended, increasing risk for maternal and infant morbidity and mortality. Most unintended pregnancies occur in the context of contraceptive non-use or failure. Women with husbands who are not supportive of contraception are more likely to report contraceptive non-use, and women with sexually abusive husbands are more likely to report contraceptive failure. This highlights the need for family planning (FP) interventions that engage both women and men, focus on eliminating marital sexual violence (MSV) and promote use of effective contraceptives including long-acting reversible contraception (LARC). Rural India, with some of the lowest rates of contraception and highest rates of marital violence globally, offers an important context to test such interventions, with global implications. Prior research from this team documents promise of the original CHARM intervention, a gender equity (GE) FP intervention engaging men and delivered by male health providers over 3 months. This intervention improved contraceptive use and reduced likelihood of MSV, but demonstrated no reduction in unintended pregnancy; additionally, it demonstrated high participation from men (91%) but less from couples (51%), largely due to women's discomfort with a male provider. Poor reach to women and provision of only short-acting contraceptives, more vulnerable to contraceptive failure, may have compromised an effect on unintended pregnancy outcomes. Based on these findings, CHARM2 includes CHARM sessions for men AND parallel women-focused GE+FP sessions delivered by a female provider and inclusive of broader contraceptive options, including LARC. This study seeks a) to implement CHARM2, b) to evaluate its impact on contraceptive use, unintended pregnancy, and MSV with rural couples in India, and c) to assess its potential for sustainability in rural India, using implementation science methods.

To evaluate the impact of CHARM2, a 2-armed cluster randomized controlled trial will be conducted with up to N=1200 married couples from 20 geographic clusters (n=50-60 couples per cluster) in rural India. Participants will receive CHARM2 or the standard of care, which will involve community health workers offering pills/condoms and linking women to public health clinics. Outcomes will be assessed via pregnancy testing and surveys at baseline, 9 & 18-month follow-ups. Implementation science methods will assess the quality, scalability, and replicability of CHARM2 for uptake by rural health care systems (i.e., sustainability).

DETAILED DESCRIPTION:
Overview: This study will involve 3 phases: Phase 1- the Preparatory Phase to map the project area and prepare communities for the planned research. Phase 2- Implementation and Evaluation of CHARM 2 (Aims 1&2), using a two-armed cluster randomized controlled trial (RCT) in 20 geographic clusters mapped in Phase 1. To assess treatment impact on contraceptive use, MSV and unintended pregnancy, clusters will be randomized to receive CHARM2 or the control program, which includes standard of care public health FP services. Intervention effects will be assessed via surveys and pregnancy testing at baseline and 9 &18-month follow-up with n=1000-1200 couples (wife aged 18-29 years). Phase 3- Implementation Science Assessments will include in-depth interviews with CHARM2 providers (n=20), select CHARM2 couples (n=50) and key Indian stakeholders in FP & public health (n=50). Interviews with providers and couples will explore intervention delivery and perceived impact. Interviews with FP & public health stakeholders will obtain feedback on perceived feasibility to sustain and scale up CHARM2. A cost-effectiveness analysis will also be done to support considerations of sustainability.

Intervention: The CHARM2 intervention will involve gender, culture and contextually-tailored FP+GE counseling sessions delivered individually to husbands by a trained male health provider (2 sessions), and, in parallel, delivered individually to wives by a trained female provider (2 session2). CHARM2 differs from the original CHARM intervention by 1.) eliminating the couple session 2.) adding a parallel component for wives, delivered by a female and inclusive of reproductive coercion counseling 3.) including LARC counseling for husbands and wives and LARC provision via the public health system.

Standard of Care (Control): Under India's public health system, frontline health workers, including nurses, provide household visits to women to increase awareness and use of FP services but they rarely providing contraceptives. For those women or couples that reach the health center, standard of care FP counseling and services are delivered by a physician; free contraceptives are then offered.

Timeline: Phase 1 of the study preparation will take approximately 3 months. Phase 2 will be in month 4 to month 60, including enrollment and intervention start at month 4, 9 month follow up at month 13, and a 18 month follow up at month 22. The outcome analysis will also be carried out in this phase at month 40. Phase 3, on sustaining the intervention will overlap from month 7 to month 60.

Plan for Data Collection: All survey data will be collected using mobile devices (tablets) with an ODK-based software system for e-data collection and web-based data management. The ODK application with CHARM2 survey questionnaire will be loaded onto the tablets, displaying questions simultaneously in English and Marathi.

ELIGIBILITY:
Inclusion Criteria:

* Young wives (aged 18 - 29 years) and their husbands
* Couples fluent in Marathi and both willing to participate
* No sterilization or infertility (infertility is defined as having no pregnancy for 1+ years despite non-use of traditional or modern contraception)
* No pregnancy or female/male surgical sterilization planned for the next 18 months
* Residing in the village for at least 2 years and residing together for at least 3 months, to facilitate follow-up tracking

Exclusion Criteria

- If either member of the couple appears to be cognitively impaired or of too poor health to be able to respond to the screening assessment across 2 visits one week apart, the couple will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2402 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anita Raj, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- Junnar Taluka, Pune District, Maharashtra, India

REFERENCES:
- [Background] Raj A, Ghule M, Ritter J, Battala M, Gajanan V, Nair S, Dasgupta A, Silverman JG, Balaiah D, Saggurti N. Cluster Randomized Controlled Trial Evaluation of a Gender Equity and Family Planning Intervention for Married Men and Couples in Rural India. PLoS One. 2016 May 11;11(5):e0153190. doi: 10.1371/journal.pone.0153190. eCollection 2016. PMID 27167981
- [Background] Yore J, Dasgupta A, Ghule M, Battala M, Nair S, Silverman J, Saggurti N, Balaiah D, Raj A. CHARM, a gender equity and family planning intervention for men and couples in rural India: protocol for the cluster randomized controlled trial evaluation. Reprod Health. 2016 Feb 20;13:14. doi: 10.1186/s12978-016-0122-3. PMID 26897656
- [Background] Dixit A, Averbach S, Yore J, Kully G, Ghule M, Battala M, Begum S, Johns NE, Vaida F, Bharadwaj P, Wyss N, Saggurti N, Silverman J, Raj A. A gender synchronized family planning intervention for married couples in rural India: study protocol for the CHARM2 cluster randomized controlled trial evaluation. Reprod Health. 2019 Jun 25;16(1):88. doi: 10.1186/s12978-019-0744-3. PMID 31238954
- [Result] Johns NE, Dixit A, Ghule M, Begum S, Battala M, Kully G, Silverman J, Dehlendorf C, Raj A, Averbach S. Validation of the Interpersonal Quality of Family Planning Scale in a rural Indian setting. Contracept X. 2020 Jul 26;2:100035. doi: 10.1016/j.conx.2020.100035. eCollection 2020. PMID 32793878
- [Result] Chen GL, Silverman JG, Dixit A, Begum S, Ghule M, Battala M, Johns NE, Raj A, Averbach S. A cross-sectional analysis of intimate partner violence and family planning use in rural India. EClinicalMedicine. 2020 Apr 18;21:100318. doi: 10.1016/j.eclinm.2020.100318. eCollection 2020 Apr. PMID 32322807
- [Result] Raj A, Ghule M, Johns NE, Battala M, Begum S, Dixit A, Vaida F, Saggurti N, Silverman JG, Averbach S. Evaluation of a gender synchronized family planning intervention for married couples in rural India: The CHARM2 cluster randomized control trial. EClinicalMedicine. 2022 Mar 5;45:101334. doi: 10.1016/j.eclinm.2022.101334. eCollection 2022 Mar. PMID 35274093
- [Derived] Averbach S, Johns NE, Tomar S, Meurice ME, Rao N, Ghule M, Raj A. Psychometric evaluation of the desire to avoid pregnancy scale in India. Contraception. 2025 Aug;148:110940. doi: 10.1016/j.contraception.2025.110940. Epub 2025 May 8. PMID 40348316
- [Derived] Raj A, Johns N, Vaida F, Ghule M, Rao N, Silverman JG. Four-year follow-up of CHARM2, an effective family planning intervention, on number and sex of births: Findings from an RCT in rural India. Dialogues Health. 2025 Apr 19;6:100218. doi: 10.1016/j.dialog.2025.100218. eCollection 2025 Jun. PMID 40342544
- [Derived] Averbach S, Johns NE, Ghule M, Dixit A, Begum S, Battala M, Saggurti N, Silverman J, Raj A. Understanding quality of contraceptive counseling in the CHARM2 gender-equity focused family planning intervention: Findings from a cluster randomized controlled trial among couples in rural India. Contraception. 2023 Feb;118:109907. doi: 10.1016/j.contraception.2022.10.009. Epub 2022 Nov 1. PMID 36328094
- [Derived] Dixit A, Johns NE, Ghule M, Battala M, Begum S, Yore J, Saggurti N, Silverman JG, Reed E, Benmarhnia T, Averbach S, Raj A. Male-female concordance in reported involvement of women in contraceptive decision-making and its association with modern contraceptive use among couples in rural Maharashtra, India. Reprod Health. 2021 Jun 30;18(1):139. doi: 10.1186/s12978-021-01187-8. PMID 34193214

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study involves randomization at the geographic cluster level. Clusters were created based on geographic boundaries surrounding a subcenter health facility. Clusters were randomized to intervention or control conditions using computer-generated random numbers. Households within each cluster were screened sequentially for eligibility. The required number of couples per cluster (n=60) were selected through systematic random sampling (selecting every nth participant).
Units Other Than Participants: Subcenters (geographic catchment areas)
Period: Overall Study
Arm/Group | CHARM2 Intervention | Control
Started | 1200; 10 Subcenters (geographic catchment areas) | 1202; 10 Subcenters (geographic catchment areas)
9 Month Follow-up | 1091; 10 Subcenters (geographic catchment areas) | 1114; 10 Subcenters (geographic catchment areas)
Completed | 1080; 10 Subcenters (geographic catchment areas) | 1110; 10 Subcenters (geographic catchment areas)
Not Completed | 120; 0 Subcenters (geographic catchment areas) | 92; 0 Subcenters (geographic catchment areas)
Not completed — Death | 3 | 3
Not completed — Lost to Follow-up | 117 | 89

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CHARM2 Intervention | Control | Total
Number analyzed (Participants) | 1200 | 1202 | 2402
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1200 | 1202 | 2402
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 600 | 601 | 1201
  Male | 600 | 601 | 1201
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1200 | 1202 | 2402
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  India | 1200 | 1202 | 2402

OUTCOME MEASURES:

1. Primary Outcome: Number of Non-pregnant Couples With Modern Contraceptive Use in Past 3 Months
Description: Based on self-report in survey on item assessing form of contraceptive used in past 3 months, with all types of traditional and modern contraceptives included as options. Variable will be constructed by dichotomizing data as yes/no for use of modern contraceptives. This measure was taken from the Demographic and Health Survey (DHS) and has been used in India's DHS for decades.
  This outcome excludes currently pregnant couples.
Time Frame: 18 months
Population: This outcome is analyzed at the couple level, based on wife report (wife report has been shown to be most reliable). This outcome includes only non-pregnant couples. Pregnant couples are excluded from this outcome. The outcome is also missing if only husband provided survey data at 18 months (N=9 intervention, N=6 control)
Measure: Count of Units; unit: Couple
Units Other Than Participants: Couple
Arm/Group | CHARM2 Intervention | Control
Number analyzed (Participants) | 998 | 1012
Number analyzed (Couple) | 499 | 506
Couple | 265 | 295

2. Secondary Outcome: Number of Couples Reporting Marital Sexual Violence
Description: Marital Sexual Violence will be assessed via two items asked of wives on forced or pressured sexual activity from husband in the past six months, dichotomized based on a yes response to either item. These items were taken from the Demographic and Health Survey. Prior research from India documents a Cronbach's alpha for this two item measure of 0.97.
Time Frame: 18 months
Population: This outcome is analyzed at the couple level as it relies on wife's report. The outcome is missing if only the husband provided 18-month survey data (N=9 intervention, N=6 control).
Measure: Count of Units; unit: Couples
Units Other Than Participants: Couples
Arm/Group | CHARM2 Intervention | Control
Number analyzed (Participants) | 1072 | 1104
Number analyzed (Couples) | 536 | 552
Couples | 7 | 5

3. Secondary Outcome: Number of Couples Reporting Unintended Pregnancy During Follow-up Time Period
Description: This outcome will be constructed based on reported pregnancy during the 18-month follow up time period, and a question asked of the female participant in reference to each pregnancy whether they had wanted the pregnancy at that time, not at that time but in the future, or not at all. If participants indicate that they did not want at least one pregnancy during the follow-up time period at that time or at all, they were be identified as having an unintended pregnancy.
Time Frame: 18 months
Population: This outcome is analyzed at the couple level as it relies on wife's report. It includes N=11 intervention couples and N=7 control couples where the wife provided information at 9-month follow-up but not 18-month follow-up. It is missing for N=25 intervention couples and N=25 control couples where the wife declined or was missing information on pregnancy intendedness.
Measure: Count of Units; unit: Couple
Units Other Than Participants: Couple
Arm/Group | CHARM2 Intervention | Control
Number analyzed (Participants) | 1044 | 1068
Number analyzed (Couple) | 522 | 534
Couple | 58 | 69

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | CHARM2 Intervention | Control
All-Cause Mortality (participants affected / at risk) | 3/1200 | 3/1202
Serious Adverse Events (participants affected / at risk) | 0/1200 | 0/1202
Other Adverse Events (participants affected / at risk) | 0/1200 | 0/1202

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/14/NCT03514914/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/14/NCT03514914/ICF_001.pdf